CLINICAL TRIAL: NCT03375463
Title: Pharmacokinetics, Safety, and Tolerability of a Solution Formulation of LY3298176 in Healthy Subjects
Brief Title: A Study of Tirzepatide (LY3298176) in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 16671; I8F-MC-GPGE (Other: Eli Lilly and Company)
Record Dates: First submitted 2017-12-13; First posted 2017-12-18 (Actual); Results first posted 2024-02-05 (Actual); Last update posted 2024-02-05 (Actual); Status verified 2024-02

CONDITIONS: Healthy
MeSH Terms: interventions — Tirzepatide

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Part A, B and D are not blinded. Part C is blinded to Participant and Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- 5 mg Tirzepatide SC (Solution)-Part A (Experimental): Participants received 5 milligrams (mg) of tirzepatide subcutaneous (SC) solution formulation.
  Interventions: Drug: Tirzepatide
- 5 mg Tirzepatide SC (Lyophilized)-Part A (Experimental): Participants received 5 mg of tirzepatide SC lyophilized formulation.
  Interventions: Drug: Tirzepatide
- 0.5 mg LY3298176 IV-Part B (Experimental): Participants received Intravenous (IV) infusion of a single 0.5 mg dose of tirzepatide formulation.
  Interventions: Drug: Tirzepatide
- 5 mg/7.5 mg/ 10 mg Tirzepatide SC-Part C (Experimental): Participants received tirzepatide subcutaneous solution at 5 mg on Days 1 (week 1) and 8 (Week 2), 7.5 mg on Day 15 (Week 3) and 10 mg on Day 22 (Week 4).
  Interventions: Drug: Tirzepatide
- Placebo SC-Part C (Placebo Comparator): Participants received SC injection of placebo.
  Interventions: Drug: Placebo
- 0.5 mg LY3298176 Bolus IV-Part D (Experimental): Participants received IV bolus of 0.5 mg tirzepatide lyophilized formulation.
  Interventions: Drug: Tirzepatide

INTERVENTIONS:
Drug: Tirzepatide — Administered SC
  Other Names: LY3298176
  Arms: 5 mg Tirzepatide SC (Lyophilized)-Part A; 5 mg Tirzepatide SC (Solution)-Part A; 5 mg/7.5 mg/ 10 mg Tirzepatide SC-Part C
Drug: Tirzepatide — Administered IV
  Other Names: LY3298176
  Arms: 0.5 mg LY3298176 IV-Part B
Drug: Placebo — Administered SC
  Arms: Placebo SC-Part C
Drug: Tirzepatide — Administered IV
  Other Names: LY3298176
  Arms: 0.5 mg LY3298176 Bolus IV-Part D

SUMMARY:
This study has four parts. Each participant will enroll in one part.

Part A: The purpose of Part A is to compare study drug tirzepatide solution formulation to a powder formulation mixed with water and given subcutaneously (SC) (just under the skin). Part A will measure how much of the study drug gets into the blood stream and how long it takes the body to get rid of it.

Part B: The purpose of Part B is to evaluate the safety and tolerability of tirzepatide intravenous (IV) formulation when administered into a vein.

Part C: The purpose of Part C is to evaluate the safety and tolerability of tirzepatide following multiple SC weekly doses of a solution.

Part D: The purpose of Part D is to evaluate the safety and tolerability of tirzepatide following single IV bolus dose of lyophilized formulation.

This study will last approximately 70 days for each part (Part A, Part B or Part D) and 92 days for Part C. This does not include screening. Screening is required within 28 days prior to the start of the study.

ELIGIBILITY:
Inclusion Criteria:

* Overtly healthy males or females, as determined by medical history and physical examination
* Male participants: agree to use an effective method of contraception for the duration of the study and for 3 months following the last dose of investigational product
* Female participants: not of childbearing potential due to surgical sterilization (hysterectomy or bilateral oophorectomy or tubal ligation) or menopause. Women with an intact uterus are deemed postmenopausal if they are greater than or equal to (≥)45 years old and have not taken hormones or oral contraceptives within the last year and had cessation of menses for at least 1 year. Or, have had at least 6 months of amenorrhea with follicle-stimulating hormone levels consistent with a postmenopausal state
* Have a body mass index of 18.5 to 32.0 kilograms per meter squared (kg/m²) inclusive

Exclusion Criteria:

* Currently enrolled in a clinical trial involving an investigational product or any other type of medical research judged not to be scientifically or medically compatible with this study
* Received treatment with a drug that has not received regulatory approval for any indication within 30 days of screening
* Have a history of heart block, or a pulse rate (PR) interval greater than (>)200 milliseconds (msec), or any abnormality in the 12-lead electrocardiogram (ECG) at screening that, in the opinion of the investigator, increases the risks associated with participating in the study
* Have a significant history of or current cardiovascular (myocardial infarction, congestive heart failure, cerebrovascular accident, venous thromboembolism, etc.), respiratory, hepatic, renal, gastrointestinal (GI), endocrine, hematological (including history of thrombocytopenia), or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs, or of constituting a risk when taking the study medication, or interfering with the interpretation of data

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2017-12-19 (Actual); Primary Completion 2018-12-27 (Actual); Study Completion 2018-12-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- Covance, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 4-part study, Part A (2-period, 2-treatment, crossover study with at least 35 days of washout period), Part B (fixed, single-arm treatment study), Part C (placebo-controlled, 4-week dose escalation study) and Part D (a fixed, single-arm treatment study).
Groups:
- Sequence 1-Part A: Participants received 5 milligrams (mg) of tirzepatide subcutaneous (SC) solution formulation in Period 1 and 5 mg of tirzepatide SC lyophilized formulation in Period 2.
- Sequence 2-Part A: Participants received 5 mg of tirzepatide SC lyophilized formulation in Period 1 and 5 mg of tirzepatide SC solution formulation in Period 2.
- 0.5 mg Tirzepatide IV-Part B: Participants received Intravenous (IV) infusion of a single 0.5 mg dose of tirzepatide solution formulation.
- 5 mg/7.5 mg/ 10 mg Tirzepatide SC-Part C: Participants received tirzepatide subcutaneous solution formulation at 5 mg on Days 1 (week 1) and 8 (Week 2), 7.5 mg on Day 15 (Week 3) and 10 mg on Day 22 (Week 4).
- 0.5 mg Tirzepatide Bolus IV-Part D: Participants received IV bolus of 0.5 mg tirzepatide lyophilized formulation.
Period: Period 1
Arm/Group | Sequence 1-Part A | Sequence 2-Part A | 0.5 mg Tirzepatide IV-Part B | Placebo SC-Part C | 5 mg/7.5 mg/ 10 mg Tirzepatide SC-Part C | 0.5 mg Tirzepatide Bolus IV-Part D
Started | 10 | 10 | 8 | 4 | 12 | 8
Received at Least 1 Dose of Study Drug | 10 | 10 | 8 | 4 | 12 | 8
Completed | 10 | 10 | 7 | 4 | 11 | 8
Not Completed | 0 | 0 | 1 | 0 | 1 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 1 | 0
Period: Period 2
Arm/Group | Sequence 1-Part A | Sequence 2-Part A | 0.5 mg Tirzepatide IV-Part B | Placebo SC-Part C | 5 mg/7.5 mg/ 10 mg Tirzepatide SC-Part C | 0.5 mg Tirzepatide Bolus IV-Part D
Started | 10 | 10 | 0 (Part B was planned as a single Period study.) | 0 (Part C was planned as a single Period study.) | 0 (Part C was planned as a single Period study.) | 0 (Part D was planned as a single Period study.)
Received at Least 1 Dose of Study Drug | 10 | 10 | 0 | 0 | 0 | 0
Completed | 9 | 9 | 0 | 0 | 0 | 0
Not Completed | 1 | 1 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 1 | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Sequence 1-Part A | Sequence 2-Part A | 0.5 mg Tirzepatide IV-Part B | Placebo SC-Part C | 5 mg/7.5 mg/ 10 mg Tirzepatide SC-Part C | 0.5 mg Tirzepatide Bolus IV-Part D | Total
Number analyzed (Participants) | 10 | 10 | 8 | 4 | 12 | 8 | 52
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 10 | 10 | 8 | 4 | 11 | 8 | 51
  >=65 years | 0 | 0 | 0 | 0 | 1 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 0 | 0 | 7 | 4 | 15
  Male | 8 | 8 | 8 | 4 | 5 | 4 | 37
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 1 | 1 | 1 | 1 | 2 | 9
  Not Hispanic or Latino | 7 | 9 | 7 | 3 | 11 | 6 | 43
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 1 | 0 | 0 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 5 | 7 | 3 | 2 | 8 | 4 | 29
  White | 5 | 2 | 4 | 2 | 4 | 3 | 20
  More than one race | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 10 | 10 | 8 | 4 | 12 | 8 | 52

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics (PK) Part A: Area Under the Concentration Versus Time Curve [AUC (0-∞)] of Tirzepatide
Description: Pharmacokinetics (PK) Part A: Area under the concentration versus time curve [AUC (0-∞)] of tirzepatide.
Time Frame: Part A: Predose, 8, 12, 24, 48, 72, 96, 120, 144, 168, 336, 480, 816-864 hours postdose
Population: All randomized participants from Part A group, who received at least one dose of study drug and had evaluable PK data
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms*hours per milliliter(ng*hr/mL)
Groups:
- 5 mg Tirzepatide SC (Solution)-Part A: Participants received 5 mg of tirzepatide SC solution formulation.
Arm/Group | 5 mg Tirzepatide SC (Lyophilized)-Part A | 5 mg Tirzepatide SC (Solution)-Part A
Number analyzed (Participants) | 19 | 20
nanograms*hours per milliliter(ng*hr/mL) | 113000 (19) | 109000 (17)

2. Primary Outcome: PK Part A: Maximum Observed Drug Concentration (Cmax) of Tirzepatide
Description: PK Part A: Maximum observed plasma drug concentration (Cmax) of tirzepatide.
Time Frame: Part A: Predose, 8, 12, 24, 48, 72, 96, 120, 144, 168, 336, 480 and 816-864 hours postdose
Population: All randomized participants from Part A group, who received at least one dose of study drug and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per milliliter (ng/mL)
Arm/Group | 5 mg Tirzepatide SC (Lyophilized)-Part A | 5 mg Tirzepatide SC (Solution)-Part A
Number analyzed (Participants) | 20 | 20
nanograms per milliliter (ng/mL) | 524 (27) | 575 (22)

3. Primary Outcome: PK Part B: Area Under the Concentration Versus Time Curve [AUC (0-∞)] of Tirzepatide
Description: PK Part B: Area under the concentration versus time curve [AUC (0-∞)] of tirzepatide.
Time Frame: Part B: Predose, 0.08 hours (h), 0.16h, 0.5h, 1h, 2h, 4h, 8h, 12h, 24h, 36h, 48h, 72h, 96h, 120h, 144h, 168h, 336h, 816h-864h and >=70 days post dose
Population: All randomized participants from Part B group, who received at least one dose of study drug and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Groups:
- 0.5 mg Tirzepatide IV-Part B: Participants received IV infusion of a single 0.5 mg dose of tirzepatide solution formulation.
Arm/Group | 0.5 mg Tirzepatide IV-Part B
Number analyzed (Participants) | 8
ng*hr/mL | 6680 (26)

4. Secondary Outcome: PK Part C: Area Under the Concentration Versus Time Curve [AUC (0-τ)] of Tirzepatide
Description: PK Part C: Area under the concentration versus time curve during one dosing interval (168 hours) [AUC (0-τ)] of tirzepatide.
Time Frame: Part C: Predose, 8 hours (h) (day (D)1), 24h (D2), 48h (D3),72h (D4), predose (D8), predose (D15), 8h (D15), 24h (D16), 48h (D17), 72h (D18), predose (D22), 8h (D22), 24h (D23), 48h (D24), 72h (D25), D57 and >= D96 postdose
Population: All randomized participants from Part C group, who received at least one dose of study drug and had evaluable PK data. As per planned analysis, for 10 mg Tirzepatide SC-Part C arm, no PK samples were collected at 168 hour post dose (after the fourth dose. i.e. following dose at Week 4). Hence, no data was collected to calculate AUC (0-τ) for 10 mg Tirzepatide SC-Part C arm.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Groups:
- 5 mg Tirzepatide SC-Part C: Participants received 5 mg of tirzepatide subcutaneous solution formulation on day 1 (week 1).
- 7.5 mg Tirzepatide SC-Part C: Participants received 7.5 mg of tirzepatide subcutaneous solution formulation on day 15 (week 3).
- 10 mg Tirzepatide SC-Part C: Participants received 10 mg of tirzepatide subcutaneous solution formulation on day 22 (week 4).
Arm/Group | 5 mg Tirzepatide SC-Part C | 7.5 mg Tirzepatide SC-Part C | 10 mg Tirzepatide SC-Part C
Number analyzed (Participants) | 12 | 12 | 0
ng*hr/mL | 68900 (19) | 149000 (26) |

5. Secondary Outcome: PK Part C: Maximum Observed Drug Concentration (Cmax) of Tirzepatide
Description: PK Part C: Maximum observed plasma drug concentration (Cmax) of tirzepatide.
Time Frame: as for outcome 4
Population: All randomized participants participants from Part C group, who received at least one dose of study drug and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- 7.5 mg LY3298176 SC-Part C: Participants received 7.5 mg of tirzepatide subcutaneous solution formulation on day 15 (week 3).
Arm/Group | 5 mg Tirzepatide SC-Part C | 7.5 mg LY3298176 SC-Part C | 10 mg Tirzepatide SC-Part C
Number analyzed (Participants) | 12 | 12 | 11
ng/mL | 663 (23) | 1270 (24) | 1900 (24)

6. Secondary Outcome: PK Part D: Area Under the Concentration Versus Time Curve [AUC (0-∞)] of Tirzepatide
Description: PK Part D: Area under the concentration versus time curve [AUC (0-∞)] of tirzepatide.
Time Frame: Part D: Predose, 0.08 hours (h), 0.16h, 0.5h, 1h, 2h, 4h, 8h, 12h, 24h, 36h, 48h, 72h, 96h, 120h, 144h, 168h, 336h, 816-864h and >= 70 days postdose
Population: All randomized participants from Part D group, who received at least one dose of study drug and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | 0.5 mg Tirzepatide Bolus IV-Part D
Number analyzed (Participants) | 8
ng*hr/mL | 14000 (16)

ADVERSE EVENTS:
Time Frame: Up To 92 Days
Description: All randomized participants who received at least one dose of study drug
Groups:
- 5 mg Tirzepatide SC, First-Part C: Participants received 5 mg of tirzepatide subcutaneous solution formulation on day 1 (week 1).
- 5 mg Tirzepatide SC, Second Dose-Part C: Participants received 5 mg of tirzepatide subcutaneous solution formulation on day 8 (Week 2).
Arm/Group | 5 mg Tirzepatide SC (Lyophilized)-Part A | 5 mg Tirzepatide SC (Solution)-Part A | 0.5 mg Tirzepatide IV-Part B | Placebo SC-Part C | 5 mg Tirzepatide SC, First-Part C | 5 mg Tirzepatide SC, Second Dose-Part C | 7.5 mg LY3298176 SC-Part C | 10 mg Tirzepatide SC-Part C | 0.5 mg Tirzepatide Bolus IV-Part D
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20 | 0/8 | 0/4 | 0/12 | 0/12 | 0/12 | 0/11 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 0/8 | 0/4 | 0/12 | 0/12 | 0/12 | 0/11 | 0/8
Other Adverse Events (participants affected / at risk) | 9/20 | 5/20 | 1/8 | 1/4 | 4/12 | 2/12 | 6/12 | 4/11 | 3/8
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 5 mg Tirzepatide SC (Lyophilized)-Part A (N=20) | 5 mg Tirzepatide SC (Solution)-Part A (N=20) | 0.5 mg Tirzepatide IV-Part B (N=8) | Placebo SC-Part C (N=4) | 5 mg Tirzepatide SC, First-Part C (N=12) | 5 mg Tirzepatide SC, Second Dose-Part C (N=12) | 7.5 mg LY3298176 SC-Part C (N=12) | 10 mg Tirzepatide SC-Part C (N=11) | 0.5 mg Tirzepatide Bolus IV-Part D (N=8)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 4 (4) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 3 (4) | 1 (1) | 0 (0)
Odynophagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site reaction (General disorders) | 5 (6) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 3 (3) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vaginal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cold sweat (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (3):
  • Study Protocol: GPGE 05 Protocol Addenda (1) (2018-08-31): https://cdn.clinicaltrials.gov/large-docs/63/NCT03375463/Prot_000.pdf
  • Study Protocol: GPGE 05 Protocol (a) (2018-01-23): https://cdn.clinicaltrials.gov/large-docs/63/NCT03375463/Prot_001.pdf
  • Statistical Analysis Plan (2017-11-30): https://cdn.clinicaltrials.gov/large-docs/63/NCT03375463/SAP_002.pdf